CLINICAL TRIAL: NCT03632343
Title: The Pain Squad+ Smartphone App To Support Real-Time Pain Management for Adolescents With Cancer: A Randomized Controlled Trial
Brief Title: The Pain Squad+ Smartphone App To Support Real-Time Pain Management for Adolescents With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Jennifer Stinson, Senior Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 1000060765
Record Dates: First submitted 2018-08-10; First posted 2018-08-15 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Therapy-Associated Cancer
Keywords: self-management; pain; adolescents; mHealth
MeSH Terms: conditions — Neoplasms, Second Primary; Pain

STUDY DESIGN:
Intervention Model Description: This will be a multi-centre, waitlist group controlled, data analyst blinded, 3-arm parallel-group superiority randomized controlled trial (RCT) with 1:1:1 allocation. Randomization will be stratified by recruitment site to account for differences in care across sites49 with block sizes of 6 and 9 within each stratum. This trial has been designed along the pragmatic end of the pragmatic-explanatory continuum. Our approach to study eligibility criteria, intervention intensity, and participant adherence will determine intervention effect under real-world conditions.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group A (Experimental): Participants in this arm will receive the Pain Squad+ smartphone app with algorithm-driven pain management advice registered nurse (RN)-initiated pain support. Email alerts related to clinically important incoming pain reports (3 consecutive reports of pain >3/10) will be sent to the study RN who will contact the healthcare team at the participants' home center to initiate clinician-driven intervention, which may be outside of the scope of the self-management algorithm. The RN will contact the participant within 12 hours of receiving the alert, including on weekends.
  Interventions: Other: Pain Squad+ with Nurse Support
- Experimental Group B (Experimental): Participants in this arm will receive the Pain Squad+ smartphone app with algorithm-driven pain management advice but without nurse (RN)-initiated pain support.
  Interventions: Other: Pain Squad+
- Waitlist Control (No Intervention): Participants in this arm will be waitlisted to receive their choice of experimental group condition within 1 month of completing all post-study outcome measures.

INTERVENTIONS:
Other: Pain Squad+ with Nurse Support — Pain Squad+ smartphone app with algorithm-driven pain management advice registered nurse (RN)-initiated pain support. Email alerts related to clinically important incoming pain reports (3 consecutive reports of pain >3/10) will be sent to the study RN who will contact the healthcare team at the participants' home center to initiate clinician-driven intervention, which may be outside of the scope of the self-management algorithm. The RN will contact the participant within 12 hours of receiving the alert, including on weekends.
  Arms: Experimental Group A
Other: Pain Squad+ — Pain Squad+ smartphone app with algorithm-driven pain management advice without RN-initiated pain support.
  Arms: Experimental Group B

SUMMARY:
Pain negatively affects the quality of life of adolescents with cancer (AWC). It can also represent a high cost to the healthcare system and families. In response, our team has built a smartphone-based app, called Pain Squad+, which can give AWC real-time advice to manage their pain. The app uses pain diaries and personalized pain advice plus support from a registered nurse to give real-time pain management in all settings. This study will look at the impact of Pain Squad+, with or without the nurse support, on AWC health quality and healthcare costs over time.

DETAILED DESCRIPTION:
Pain negatively affects the quality of life (QOL) of adolescents with cancer (AWC), slows cancer recovery, and results in negative long-term health effects. Pain is also significant cost to the healthcare system and families. To address this problem, the study investigators have developed and used a phased-approach to test a smartphone-based app, called Pain Squad+. Using this app AWC report the pain they have and the app provides AWC with advice on how to treat this pain based on an algorithm our team developed. An email is also sent to a nurse if an AWC reports severe pain 3 times in a row. The nurse then contacts the AWC to assist in treating pain. This project will test the effect of the Pain Squad+ app, with and without nurse help, on treating pain and other pain-related health issues and managing costs associated with pain care, when compared to AWC not using the app. Investigators will enroll 222 AWC recruited from 9 Canadian pediatric oncology care centres into a 3-group randomized controlled trial. AWC in the experimental groups will be asked to use Pain Squad+ for 8 weeks (with or without nurse involvement) and all groups will complete pain-related outcome measures at baseline, 2-, 4-, 8-, and 16-weeks. The primary study outcome will be pain intensity. The secondary study outcomes will be (a) pain interference; (b) QOL; (c) pain self-efficacy; and (d) cost effectiveness and utility. Investigators will use established statistical methods to analyze the health and cost data collected over the course of this study. A real-time and cost effective way to address the problem of pain in AWC is needed. Pain Squad+ can improve pain treatment and QOL for AWC as well as decrease costs incurred by families and the healthcare system. If effective, the Pain Squad+ as a model of technology-assisted care may represent a way to improve the QOL for a range of Canadian patients by treating a variety of physical and psychological symptoms the moment they occur.

ELIGIBILITY:
Inclusion Criteria:

* aged 12-18 years,
* are able to speak and read English,
* are diagnosed with cancer (all disease types),
* are on active therapy,
* have an average self-reported pain score of ≥3/10 measured using an 11-point numerical rating scale (NRS) over the preceding week, and
* have an English-speaking and reading caregiver who is willing and able to complete outcome measures related to healthcare encounters

Exclusion Criteria:

* with significant cognitive impairments or co-morbid illnesses (as determined by their medical team) that would limit interaction with Pain Squad+ or outcome measure assessment,
* who are currently participating in other pain management studies, and
* who are not expected to survive past 16 weeks as determined by their oncologist

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 102 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) | Change from baseline Brief Pain Inventory measure at 4 time points: 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline, 16 weeks after baseline
  The BPI assesses current pain and 'worst', 'least', and 'average' pain in the preceding week using an 11-point numerical rating scale (NRS) with verbal anchors 'no pain' at 0 and 'pain as bad as you can imagine' at 10. Item scores are averaged to give a Pain Intensity Summary Score.

SECONDARY OUTCOMES:
Patient Reported Outcomes Measurement Information System (PROMIS) Pediatric Pain Interference Short-form Scale | Baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline, 16 weeks after baseline
  The PROMIS instrument is a valid 8- item scale assessing the impact of pain on function. Higher scores represent greater interference with function. We will use the established Bonferroni correction to account for serial comparisons.
Pediatric Quality of Life Inventory (PedsQL) 4.0 | Baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline, 16 weeks after baseline
  The PedsQL 4.0 is a valid and reliable 23-item instrument not specific to pain. It is comprised of 4 subscales (physical functioning, emotional functioning, social functioning and school functioning), which are summed to provide a total score. Higher scores represent better QOL. We will separately analyze the subscales and total scale scores of the PedsQL.
Porter's scale | Baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline, 16 weeks after baseline
  Porter's scale which assesses self-efficacy for managing pain, symptoms, and function in cancer patients. This 16-item scale includes a valid and reliable 5-item subscale assessing cancer pain management self-efficacy with higher scores indicating more certainty and is adapted from a scale that has been successfully administered to adolescents.
Health Utility Index Mark 2/3 (HUI2/3) | Baseline, 8 weeks after baseline, 16 weeks after baseline
  Quality-adjusted life years (QALYs)68 will be calculated using data from the valid and reliable HUI2/3.
Health Services Use | Baseline, 8 weeks after baseline, 16 weeks after baseline
  Direct healthcare costs will include the intervention and costs for health service use by AWC during the trial. Family out-of-pocket expenses, indirect costs due to lost productivity, and health service use will be ascertained using standardized customized data collection forms.

OTHER OUTCOMES:
Adolescent Demographic Questionnaire | Baseline
  This questionnaire will ask about socio-economic, demographic, and disease information for descriptive purposes. It will also obtain information on potential moderators of observed treatment effects: AWC age, sex, ethnicity, school grade, diagnosis, stage/risk, relapse-status, treatment-type, date of diagnosis, co-morbid conditions and medications, and pain history.
Parent Demographic Questionnaire | Baseline
  This questionnaire will ask about parents about their age, sex, ethnicity, educational attainment, and financial characteristics

CONTACTS AND LOCATIONS:
Locations (9):
- Canada (9):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital London Health Sciences, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jibb L, Nathan PC, Breakey V, Fernandez C, Johnston D, Lewis V, McKillop S, Patel S, Sabapathy C, Strahlendorf C, Victor JC, Moretti ME, Nguyen C, Hundert A, Cassiani C, El-Khechen Richandi G, Insull H, Hamilton R, Fang G, Kuczynski S, Stinson J. Pain Squad+ smartphone app to support real-time pain treatment for adolescents with cancer: protocol for a randomised controlled trial. BMJ Open. 2020 Mar 16;10(3):e037251. doi: 10.1136/bmjopen-2020-037251. PMID 32184315